CLINICAL TRIAL: NCT00524836
Title: A Study Evaluating the Efficacy and Safety of 5 mg Levocetirizine Oral Tablets, Once Daily Versus 10 mg Loratadine Oral Tablets, Once Daily for the Treatment of Perennial Allergic Rhinitis.
Brief Title: Efficacy and Safety of Levocetirizine Versus Loratadine for the Treatment of Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A00349
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2009-09

CONDITIONS: Rhinitis; Allergic; Perennial
Keywords: levocetirizine dihydrochloride; Xyzal tablets
MeSH Terms: conditions — Rhinitis | interventions — levocetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: levocetirizine dihydrochloride

SUMMARY:
Efficacy and Safety of Levocetirizine Versus Loratadine for the Treatment of Perennial Allergic Rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Male ore female, 16 to 60 years old (inclusive)
* two-year history of allergic rhinitis due to house dust mite

Exclusion Criteria:

* An ear, nose or throat (ENT) infection
* asthma requiring daily drug therapy other than ß2 inhaled agonists taken prn
* atopic dermatitis or urticaria requiring an antihistamine or corticosteroid treatment
* an associated ENT disease
* use of decongestants
* nasal or ocular topical treatment
* desensitivation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2003-09; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Total 5 Symptom Score (T5SS) rated by the investigator | 2 weeks

SECONDARY OUTCOMES:
Investigators global efficacy evaluation at the end of treatment; subject's rating of T5SS and individual symptoms (over the last 24 hours) over first week and the total 2 weeks treatment period; the Symptoms Score Reducing Index (SSRI). | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma